CLINICAL TRIAL: NCT01094340
Title: "Twenty-Four-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Effect of Fixed Dose Regimens of Thalidomide and Placebo on CSF and Plasma Biomarkers in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Thalidomide for Patients With Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Banner Health (Other)
Responsible Party: Principal Investigator, Brian Browne, MARWAN SABBAGH, MD Director, Banner Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01AG034155-01 (NIH)
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidoide (Other): CSF
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — fixed dose over 8 clinic visits
  Other Names: Celegene

SUMMARY:
This is a 24-week, randomized, double-blind, placebo-controlled study of the effect of thalidomide and placebo on CSF (cerebral spinal fluid) and plasma biomarkers in patients with mild to moderate Alzheimer's disease. This study will evaluate the effects of 24 weeks of treatment with Thalidomide on plasma biomarkers.

DETAILED DESCRIPTION:
A lumbar puncture will be done before treatment (baseline), and at 24 weeks to collect CSF for the quantification of biomarkers. As an exploratory effort, we will test the effects of thalidomide on the same biomarkers in the plasma and will determine if detectable changes mirror changes observed in the CSF.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a screening diagnosis of Probable Alzheimer's disease according to National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
* Subjects must have a Mini-Mental State Examination (MMSE) score of 12-26
* Subject must live at home.
* Must have a caregiver to participate in this study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Improve cognition | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Liebsack, BSN, Study Director — Banner Health
Locations (1):
- Banner Sun Health Research Institute, Sun City, Arizona, United States